CLINICAL TRIAL: NCT04476680
Title: Influence of Military Preventive Policy for reCruit Training on COVID-19 Seroconversion
Acronym: IMPACTCOVID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Centre for Defence Medicine (Other Government)
Collaborators: Leeds Beckett University (Other); Liverpool John Moores University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1070MODREC20
Record Dates: First submitted 2020-07-16; First posted 2020-07-20 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: SARS-CoV Infection; Vitamin D Deficiency; Covid19; Acute Respiratory Tract Infection
Keywords: SARS-CoV-2; Cholecalciferol; Vitamin D Status; COVID-19; Acute Respiratory Tract Infection
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; Vitamin D Deficiency; COVID-19 | interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: Observational study in two cohorts, matched for age and latitude. One group will be taking vitamin D supplements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Military recruits (Active Comparator): Vitamin D supplementation (1000 IU/day D3 for 4 weeks, and 400 IU/d D3 as a maintenance dose)
  Interventions: Dietary Supplement: Vitamin D
- No intervention (No Intervention)

INTERVENTIONS:
Dietary Supplement: Vitamin D — Pure Encapsulations' manufacturing facility is a US Food and Drug Administration (FDA) inspected and NSF International Good Manufacturing Practices registered company.
  Other Names: Pure Encapsulations, Sudbury, MA, USA
  Arms: Military recruits

SUMMARY:
This study is intended to address the association between vitamin D status and seroconversion to SARS-CoV-2 in healthy young adults.

The primary aim of the study is to determine the rates of 'silent' seroconversion rates, consistent with asymptomatic transmission of SARS-CoV-2, in a young healthy adult population with a wide spread of vitamin D concentrations.

The secondary aims of this study are to explore:

1. Any effect of vitamin D status on symptomatic illness.
2. The background 'point' prevalence and subsequent rate of increase in seropositivity for SARS-CoV-2 in healthy young adults.
3. The individual reductions in seropositivity to SARS-CoV-2 over time, and changes in seropositivity in a defined young adult population over time.
4. Where salivary Immunoglobulin A (IgA) may be used to provide an alternative/ complementary serological method
5. The effect (if any) of vitamin D supplementation on seroconversion rates stratified by: i) level of baseline vitamin D 'deficiency/ insufficiency/ sufficiency' status; ii) extent of BMI-defined normal/overweight/obesity cut-offs and iii) gender.

DETAILED DESCRIPTION:
The primary aim of the study is to determine the rates of 'silent' seroconversion rates, consistent with asymptomatic transmission of SARS-CoV-2, in a young healthy adult population with a wide spread of vitamin D concentrations.

The study will be conducted over 16 weeks in two populations: Service Personnel undertaking initial military training, who are supplementing with vitamin D (1000 IU/day D3 for 4 weeks, and 400 IU/d D3 as a maintenance dose), and civilian students who are not supplementing.

We will recruit adults aged 18-30 years old. Military and civilian participants will be recruited respectively in Catterick and Leeds, UK to start in coincidence with the recommencement of Autumn semester.

In accordance with our power calculation and anticipated drop-out rate, 450 volunteers will be recruited in each group. Data collected at baseline and after 5, 9, 12 and 16 weeks will include seroconversion status assessed from a validated Dried Blood Spot (DBS) method in conjunction with novel salivary antibody testing, plus structured questionnaire responses screening for Covid-19 symptoms. Physical and demographic characteristics and serum levels of vitamin D concentrations collected from participants at study entry will facilitate secondary aims in relation to exploring the influence of gender, ethnicity, body mass and body mass index (BMI) on asymptomatic seroconversion, as well as interactions with vitamin D status and supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Able to access the study sites at Leeds Beckett University's Headingley or City campuses, UK OR recruit at Infantry Training Centre, Catterick Garrison, UK
* In possession of an internet-enabled smart phone capable of receiving and responding to smartphone alerts.

Exclusion Criteria:

* Previously diagnosed with COVID-19 either by RT-PCR or serologically (either prior to the study or at initial baseline testing).
* Use of over-the-counter or prescribed vitamin D supplements currently or in the past month
* Condition conferring 'very high risk' or 'high risk' of severe COVID-19

  * have had an organ transplant
  * are having chemotherapy or antibody treatment for cancer, including immunotherapy
  * are having an intense course of radiotherapy (radical radiotherapy) for lung cancer
  * are having targeted cancer treatments that can affect the immune system (such as protein kinase inhibitors or PARP inhibitors)
  * have blood or bone marrow cancer (such as leukaemia, lymphoma or myeloma)
  * have had a bone marrow or stem cell transplant in the past 6 months, or are still taking immunosuppressant medicine
  * are pregnant or intent on becoming pregnant during the anticipated study period
  * have a learning disability
  * have a lung condition (such as cystic fibrosis, asthma, COPD, emphysema or bronchitis)
  * have heart disease (such as heart failure)
  * have high blood pressure (hypertension)
  * have diabetes
  * have chronic kidney disease
  * have liver disease (such as hepatitis)
  * have a condition affecting the brain or nerves (such as Parkinson's disease, motor neurone disease, multiple sclerosis, or cerebral palsy)
  * have a problem with the spleen or have had the spleen removed
  * have a condition with high risk of getting infections (such as SCID, sickle cell, HIV, lupus or scleroderma)
  * are taking medicine that can affect the immune system (such as steroids)
  * are very obese (a BMI of 40 or above)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 900 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-04-28 (Estimated); Study Completion 2021-04-28 (Estimated)

PRIMARY OUTCOMES:
Seroconversion | 24 weeks
  asymptomatic seroconversion for SARS-CoV-2
Interim analysis - seropositivity at 12 weeks | 12 weeks
  asymptomatic seroconversion for SARS-CoV-2

SECONDARY OUTCOMES:
Dried Blood Spot performance | 24 weeks
  Sensitivity and specificity of dried blood spot assay compared with venous blood serology
Salivary IgA performance | 24 weeks
  Sensitivity and specificity of salivary IgA compared with venous blood serology
Prevalence of SARS-CoV-2 | 24 weeks
  The background 'point' prevalence and subsequent rate of increase in seropositivity for SARS-CoV-2 in healthy young adults.
Change in seropositivity | 24 weeks
  The individual reductions in seropositivity to SARS-CoV-2 over time, and changes in seropositivity in a defined young adult population over time
Change in seroconversion rate | 24 weeks
  The effect of vitamin D supplementation on seroconversion rates stratified by: i) level of baseline vitamin D 'deficiency/ insufficiency/ sufficiency' status; ii) extent of BMI-defined normal/overweight/obesity cut-offs, iii) gender iv) ethnicity

CONTACTS AND LOCATIONS:
Overall Officials: David R Woods, MD, Study Chair — Royal Centre of Defence Medicine, Birmingham, UK; Julie P Greeves, PhD, Principal Investigator — Army Health and Performance Research, Andover, UK; Neil Walsh, PhD, Principal Investigator — Liverpool John Moores University
Locations (2):
- United Kingdom (2):
  - Headingley and City campuses, Leeds Beckett University, Leeds, Yorkshire
  - Infantry Training Centre Catterick, Catterick Garrison

IPD SHARING:
Plan to Share IPD: No
Anonymised IPD may be available upon request